CLINICAL TRIAL: NCT00333060
Title: Phase 2 Study of OT-551 Ophthalmic Solution to Prevent or Delay Progression of Nuclear Cataract Formation In Post-Vitrectomy Patients
Brief Title: Study of OT-551 Eye Drops to Prevent or Delay Progression of Nuclear Cataracts Following Vitreous Removal
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Othera Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: OT-551-002
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Epiretinal Membrane; Macular Hole
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations

INTERVENTIONS:
Drug: OT-551 ophthalmic solution

SUMMARY:
The purpose of this trial is to compare the ability of two doses of OT-551 ophthalmic solution and drug-free solution to safely and effectively prevent or delay the progression of nuclear cataracts that frequently develop as a result of vitrectomy (surgery for retina repair), thereby avoiding the need for a second surgery (cataract removal). Victrectomies involve removal of the jelly-like substance (vitreous) that is located in a cavity behind the lens.

ELIGIBILITY:
Inclusion Criteria:

* Imminent vitrectomy to repair macular holes or puckers
* Ability to be screened for eligibility and begin dosing 7-10 days in advance of the surgery
* Best corrected ETDRS visual acuity equivalent to Snellen 20/400 or better in the surgical eye and 20/100 or better in the fellow eye

Exclusion Criteria:

* Artificial lens or no lens in the surgical eye
* Cataract (greater than slight opacity or thickness) in the surgical eye
* Any other retinal abnormality which may be vision-threatening
* Serious heart, kidney, or liver disease
* Recent ophthalmic surgery (within 6 months) or ocular infection (within 30 days)
* Poorly controlled diabetes or unstable glaucoma

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2005-11; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
change in visual acuity
change in lens opacity

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Peoria, Arizona
  - Beverly Hills, California
  - Sacramento, California
  - Denver, Colorado
  - Miami, Florida
  - Tallahassee, Florida
  - Chicago, Illinois
  - Joliet, Illinois
  - Baltimore, Maryland
  - Cherry Hill, New Jersey
  - Forrest Hills, New Jersey
  - New York, New York
  - Cleveland, Ohio
  - Bala-Cynwyd, Pennsylvania
  - West Chester, Pennsylvania
  - Abilene, Texas